CLINICAL TRIAL: NCT06817616
Title: Arthroscopic Rotator Cuff Repair with Umbilical Cord-derived Mesenchymal Stem Cells for Large to Massive Rotator Cuff Tears
Brief Title: Arthroscopic Rotator Cuff Repair with UC-MSCs for Large to Massive Tears
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Woong Kyo Jeong, PI, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUAH-25-01
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Rotator Cuff Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients diagnosed with Full-Thickness Rotator Cuff Tears, Including Massive and Large Tears (Experimental)
  Interventions: Biological: Injection allogenic Umbilical Cord-derived Mesenchymal Stem Cell

INTERVENTIONS:
Biological: Injection allogenic Umbilical Cord-derived Mesenchymal Stem Cell — Biological: Allogenic Umbilical Cord - derived Mesenchymal Stem Cell
  1. Injection dosage and volume of the study drugs:
     * Low dose: 2.5X10 cells/0.5mL
  2. Number of injections: Only once during the study period
  3. Device: Ultrasound
  4. Injection technique: Injection into the lesion by investigator
  Biological: Allogenic Umbilical Cord - derived Mesenchymal Stem Cell
  1. Injection dosage and volume of the study drugs:
     - High dose: 5X10 cells/1mL
  2. Number of injections: Only once during the study period
  3. Device: Ultrasound
  4. Injection technique: Injection into the lesion by investigator

SUMMARY:
Safety Analysis of Allogeneic Umbilical Cord-Derived Mesenchymal Stem Cells in Patients Undergoing Rotator Cuff Repair for Massive or Large Rotator Cuff Tears

ELIGIBILITY:
Inclusion Criteria:

* Male or female 19 years of age and older
* Unilateral shoulder pain with a pain score of 4 or higher.
* patients with a symptom duration of at least three months who have not responded to conventional treatments, including analgesics.
* patients diagnosed with massive or extensive full-thickness rotator cuff tears confirmed by computed tomography arthrography or magnetic resonance imaging.

Exclusion Criteria:

* patients diagnosed with small or medium full-thickness rotator cuff tears among study participants with full-thickness rotator cuff tears.
* patients who have received subacromial injection therapy in the affected shoulder within the past three months.
* patients who have undergone rotator cuff surgery on the affected shoulder within the past six months.
* patients exhibiting or suspected of having the following radiological findings: malignant tumors, severe glenohumeral osteoarthritis, or bony abnormalities causing subacromial space narrowing.
* patients presenting with symptomatic cervical spine disorders.
* patients experiencing bilateral shoulder pain.
* patients diagnosed with multiple arthritis, infectious arthritis, rheumatoid arthritis, or fibromyalgia.
* patients with neurological deficits.
* Pregnant or breastfeeding patients
* patients unwilling to use effective contraception during the study period.
* patients currently infected with HBV, HCV, or HIV, or those with a positive RPR test result.
* patients with severe conditions that may affect the study, including cardiovascular diseases, renal diseases, hepatic diseases, endocrine disorders, or malignancies.
* patients who are unable to comprehend the questionnaires used for study assessments, including the Visual Analog Scale (VAS), or those with communication difficulties due to psychiatric disorders.
* Any other cases deemed inappropriate for study participation by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) pain in motion | 12 months
  Using a ruler, the score is determined by measuring the distance (mm) on the 100mm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Changes in the size of rotator cuff tears determined by MRI | 12 months
Adverse event | 12 months

OTHER OUTCOMES:
Shoulder ROM (Forward flexion, Abduction, External rotation & Internal rotation at 0 degree) | 12 months
Muscle strength (lb) | 12 months
  The strength the supraspinatus, infraspinatus,and subscapularis was measured using a handheld electronic scale
Pulse rate (beats per minute) | 12 months
  To determine the overall safety of Autologous Adipose Tissue Derived Mesenchymal Stem Cells carrier using pulse rate
Blood Pressure (mmHg) | 12 months
  To determine the overall safety of Autologous Adipose Tissue Derived Mesenchymal Stem Cells carrier using blood pressure
CBC(complete blood count) | 12 months
  The measures are composite.
Usage amount of rescue medication | 12 months
  The total dosage of rescue medication administered to participants during the study period is measured to evaluate the amount of medication required to manage symptoms after treatment.
Frequency of rescue medication | 12 months
  The frequency of rescue medication usage is measured to assess how often participants required additional medication to manage symptoms during the study period.
Blood Glucose | 12 months
  Blood glucose levels are measured to assess glycemic control and detect hyperglycemia or hypoglycemia.
BUN/Creatinine Ratio | 12 months
  The ratio of blood urea nitrogen (BUN) to creatinine is measured to evaluate kidney function.
Serum Total Protein | 12 months
  Serum total protein levels are measured to evaluate overall protein status
Serum Albumin | 12 months
  Serum albumin levels are measured to assess liver function, nutritional status, and oncotic pressure regulation.
Serum total bilirubin | 12 months
  Serum total bilirubin levels are measured to evaluate liver function
Aspartate Transaminase/Alanine Transaminase(AST/ALT) | 12 months
  AST and ALT levels are measured to assess liver function
Serum Alkaline Phosphatase(ALP) | 12 months
  Serum ALP levels are measured to evaluate liver and bone health.
Serum Gamma-Glutamyl Transferase(γ-GTP) | 12 months
  Serum γ-GTP levels are measured to assess liver function
Serum creatine kinase(CK) | 12 months
  Serum creatine kinase levels are measured to assess muscle injury
Erythrocyte Sedimentation Rate(ESR) | 12 months
  ESR is measured to assess inflammation or detect inflammatory conditions
C-Reactive Protein(CRP) | 12 months
  Serum CRP levels are measured to evaluate acute inflammation
Urine pH Levels | 12 months
  Urine pH is measured to assess acidity or alkalinity of the urine. Lower values indicate increased acidity, while higher values indicate increased alkalinity. Normal range is typically 4.5-8.0.
Urine Specific Gravity | 12 months
  Urine specific gravity is measured to evaluate urine concentration or dilution. A value closer to 1.000 indicates more diluted urine, while higher values suggest more concentrated urine. protein
Urine Protein | 12 months
  Urine protein levels are measured to assess the presence of proteinuria. Normal range is typically negative or <20 mg/dL.
Urine Glucose | 12 months
  Urine glucose levels are measured to detect glycosuria. Normal range is negative.
Urine Bilirubin | 12 months
  Urine bilirubin levels are measured to assess liver function. Normal range is negative.
Urine Blood | 12 months
  Urine blood levels are measured to detect hematuria. Normal range is negative
Urine Ketone | 12 months
  Urine ketone levels are measured to detect ketonuria. Normal range is negative
Microscopic Analysis | 12 months
  Microscopic analysis of urine is performed to identify the presence of red blood cells (RBCs), white blood cells (WBCs), crystals, casts, or bacteria, which may indicate infection, inflammation, or other pathological conditions.
Number of participants with treatment-related adverse events as assessed by NCI - CTCAE v4.0 | 12 months
  all adverse and unintended signs (including abnormal laboratory test results), symptoms, or diseases that occur in research subjects who have been administered the investigational drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anamh Hospital, Seoul, Korea, South Korea